CLINICAL TRIAL: NCT02724527
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of N91115 for Efficacy and Safety in Patients With CF Heterozygous for F508del-CFTR + Gating Mutation Being Treated With Ivacaftor
Brief Title: Study of Cavosonstat (N91115) in CF Patients Who Are Heterozygous for F508del-CFTR and a Gating Mutation and Being Treated With Ivacaftor
Acronym: SNO-7
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N91115-2CF-06
Record Dates: First submitted 2016-03-11; First posted 2016-03-31 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; N91115; Cavosonstat
MeSH Terms: conditions — Cystic Fibrosis | interventions — cavosonstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching capsule (BID administration Q12H)
  Interventions: Drug: Placebo
- Cavosonstat (N91115) 400 mg (Experimental): Cavosonstat (N91115) at 400 mg dose (100 mg x 4 capsules) (BID administration Q12H)
  Interventions: Drug: Cavosonstat

INTERVENTIONS:
Drug: Cavosonstat — CFTR modulator that stabilizes CFTR
  Other Names: N91115
  Arms: Cavosonstat (N91115) 400 mg
Drug: Placebo — Matched Placebo capsule
  Other Names: Control
  Arms: Placebo

SUMMARY:
Cavosonstat (N91115) is being studied as a potential novel therapy for cystic fibrosis (CF), and this study assesses a target population of patients who are heterozygous for F508del-CFTR and a gating mutation that is approved for treatment with ivacaftor (G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, or S549R).

DETAILED DESCRIPTION:
Assess the effect of Cavosonstat (N91115) on lung function when added to preexisting treatment with ivacaftor in adult patients with CF who are heterozygous for F508del-CFTR and a gating mutation that is approved for treatment with ivacaftor (G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, or S549R).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF, heterozygous for F508del-CFTR and a gating mutation that is approved for treatment with ivacaftor (G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, or S549R)
* Have been treated with chronic ivacaftor twice daily for at least 6 months prior to Screening (date of consent) and are currently being treated with commercially available Ivacaftor
* Negative serum pregnancy test
* Weight ≥ 40 kg at screening
* Oxygen saturation by pulse oximetry ≥ 90% breathing ambient air, at screening

Exclusion Criteria:

* Any acute infection, including acute upper or lower respiratory infections and pulmonary exacerbations that require treatment that has completed within 2 weeks of Study Day 1 or hospitalization discharge within 2 weeks of Study Day 1
* Recent infection (per investigator discretion) with organisms associated with more rapid decline in pulmonary status, for example: Burkholderia cenocepacia, Burkholderia dolosa, and Mycobacterium abscessus
* Any change in the regimen for chronic therapies for CF lung disease (e.g., Pulmozyme®, hypertonic saline, Azithromycin, TOBI®, Cayston®) within 4 weeks of Study Day 1
* Blood hemoglobin < 10 g/dL at screening
* Serum albumin < 2.5 g/dL at screening
* Abnormal liver or renal function
* History of ventricular tachycardia or other clinically significant ventricular arrhythmias
* History, including the screening assessment, of prolonged QT and/or QTcF (Fridericia's correction) interval (> 450 msec for men; > 470 msec for women)
* History of solid organ or hematological transplantation
* History of alcohol abuse or drug abuse (including cannabis, cocaine, and opioids) in the year prior to screening
* Use of continuous (24 hr/day) or nocturnal supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
The absolute change in ppFEV1 in the N91115 treated group | Baseline, week 4 and 8 assessments
  Forced Expiratory Volume (FEV) absolute measurements comparing baseline to after 4 and 8 weeks of N91115 treatment. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. ppFEV1 (predicted for age, gender, and height) is calculated using the Hankinson method.

SECONDARY OUTCOMES:
The relative change from study baseline within the active treatment group in ppFEV1 values | Baseline, week 4 and 8 assessments
  Forced Expiratory Volume relative measurements comparing baseline to after 4 and 8 weeks of N91115 treatment. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. ppFEV1 (predicted for age, gender, and height) is calculated using the Hankinson method.
Absolute change from study baseline within the active treatment group in sweat chloride | Baseline, week 4 and 8 assessments
  Sweat chloride concentration measured by pilocarpine iontophoresis, a standard clinical laboratory technique. Sweat collection accomplished with the Wescor Macroduct System.
Changes in the respiratory domain of the Cystic Fibrosis Questionnaire - Revised, (CFQ-R) | Baseline, week 4 and 8 assessments
  Patient questionnaires will compare baseline scores on their respiratory symptoms to weeks 4 and 8
Absolute change from baseline within the active treatment group in Patient Global Impression of Change | Baseline, week 4 and 8 assessments
  Patient questionnaires will compare baseline global impression of changes in health from baseline to weeks 4 and 8
Safety as determined by adverse events assessment | Baseline to 8 weeks treatment with a 28-day follow up period
  Assessments of clinical laboratory values, electrocardiogram (ECG), pulmonary exacerbations, and vital signs
Pharmacokinetic Assessment of Maximum Plasma Concentration [Cmax] for N91115 & ivacaftor | Weeks 1, 4 and 8
  Plasma collection for assessment of N91115 and ivacaftor Cmax
Pharmacokinetic Assessment of area under the plasma concentration verse time curve [AUC] for N91115 & ivacaftor | Weeks 1, 4 and 8
  Plasma collection for assessment of N91115 and ivacaftor AUC

CONTACTS AND LOCATIONS:
Overall Officials: James Chmiel, MD, Principal Investigator — Rainbow Babies and Children's Hospital/ University
Locations (12):
- United States (12):
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital - Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Medical Center of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No